CLINICAL TRIAL: NCT01921374
Title: Profile of Mother-caregivers of Children With Duchenne Muscular Dystrophy
Brief Title: Mother-caregivers of Children With Duchenne Muscular Dystrophy
Acronym: DMDK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monica Levy Andersen (Other)
Responsible Party: Sponsor-Investigator, Monica Levy Andersen, Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: DMDK
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Other Diseases or Conditions
Keywords: Duchenne;; mothers caregivers;; sleep;; hormonal profile;; cardiac profile;; biochemical profile;; inflammatory profile.
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Insulin; Hydrocortisone; Luteinizing Hormone; Follicle Stimulating Hormone; Testosterone; Estradiol; Progesterone; Vitamin B 12; Adrenocorticotropic Hormone; C-Reactive Protein; Polymerase Chain Reaction; Immunoglobulin A; Immunoglobulin G; Immunoglobulin M; Complement C3; Complement C4; Interleukin-6; Interleukin-10; Interleukin-2; Interleukin-4; Interleukin-8; Interferon-gamma; Endothelins; Dinoprostone; Intercellular Adhesion Molecule-1; Vascular Cell Adhesion Molecule-1; Tumor Necrosis Factor-alpha; Adiponectin; Leptin; Cysteine; Homocysteine; Myoglobin; Tnni3k protein, mouse; Creatine Kinase; Creatine Kinase, MB Form; Metabolome; Glucose; Cholesterol; Triglycerides; Uric Acid; Creatinine; Urea; Sodium; Potassium; Blood Sedimentation; 5-nitro-2-(3-phenylpropylamino)benzoic acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- sleep parameters (Experimental): To assess the sleep parameters.
  Interventions: Biological: sleep parameters
- cardiovascular parameters (Other): To assess the cardiovascular profile of control mothers and caregivers-mothers.
  Interventions: Biological: Cardiovascular profile
- imflammatory and immunological profile (Experimental): To assess the inflammatory profile of caregivers-mothers and control mothers
  Interventions: Biological: Inflammatory profile
- hormonal profile (Experimental): To assess the hormonal profile of caregivers-mothers and control mothers.
  Interventions: Biological: Hormonal profile
- metabolic profile (Experimental): To assess the health profile of caregivers-mothers and control mothers.
  Interventions: Biological: Metabolic profile

INTERVENTIONS:
Biological: sleep parameters — Since the mother-caregiver dedicates herself entirely to her son, we will performe overnight polysomnography to assess the sleep pattern.
  Arms: sleep parameters
Biological: Hormonal profile — To assess the health profile of caregivers-mothers are analyzed some markers that may indicate an impairment or damage to the health of each of the parameters.
  Other Names: Insulin; Cortisol; Luteinizing hormone (LH); Follicle-stimulating hormone (FSH); Total Testosterone; Estradiol; Progesterone; Vitamin B12; Adrenocorticotropic hormone (ACTH)
  Arms: hormonal profile
Biological: Inflammatory profile — To assess the health profile of caregivers-mothers are analyzed some markers that may indicate an impairment or damage to the health of each of the parameters
  Other Names: C-reactive protein (PCR); Immunoglobulin A (IgA); Immunoglobulin G (IgG); Immunoglobulin M (IgM); Complement (C3); Complement (C4); Interleukin 6; Interleukin 10; Interleukin 1β; Interleukin 2; Interleukin 4; Interleukin 8; Interferon-gamma (IFN-γ); Endothelin; Prostaglandin E2; Intercellular Adhesion Molecule 1 (ICAM); Vascular cell adhesion protein 1 (VCAM); Tumor necrosis factor (TNFα); Adiponectin; Leptin; Cysteine; Lymphocytes subpopulations (T e B)
  Arms: imflammatory and immunological profile
Biological: Cardiovascular profile — To assess the health profile of caregivers-mothers are analyzed some markers that may indicate an impairment or damage to the health of each of the parameters
  Other Names: Homocysteine; Myoglobin; Cardiac troponin I; Creatine kinase (CK); Creatine kinase MB (CKMB)
  Arms: cardiovascular parameters
Biological: Metabolic profile — To assess the health profile of caregivers-mothers are analyzed some markers that may indicate an impairment or damage to the health of each of the parameters
  Other Names: Glucose; Total cholesterol and fractions; Triglycerides; Uric acid; Creatinine; Urea; Sodium; Potassium; Hemogram; Erythrocyte sedimentation rate; Natriuretic Peptide B
  Arms: metabolic profile

SUMMARY:
The incidence of Duchenne Muscular Dystrophy (DMD) is approximately 1 in 3.500 male newborns. During its progression there is loss of mobility, swallowing difficulties and a significant reduction in respiratory capacity. Due to the severity and consequences, is inevitable the need for a caregiver, that normally rely the mother.

DETAILED DESCRIPTION:
The Duchenne Muscular Dystrophy (DMD) is a neuromuscular disease characterized by genetic alteration, whose consequence is the progression of muscle degeneration. The mother-caregiver dedicates herself entirely to her son, putting aside the care of their physical and psychological health. The responsibility and workload to care for the child is high. Because of this extreme amount of work associated with other factors such as stress, this mothers-caregivers are more likely to develop hypertension, respiratory disease, susceptibility to infections, depression, anxiety, insomnia, impaired immune and cardiovascular problems. Moreover, they are more likely to develop sleep disorders, those who may cause a high health risk, since many sleep disorders are related to cardiovascular, respiratory, neurological and immune systems.

ELIGIBILITY:
Inclusion Criteria:

* Mothers-caregivers of children and adolescents with DMD
* Mothers of children and adolescents without any neuromuscular disease and that does not have any chronic disease (bronchiolitis obliterates, cystic fibrosis, a genetic syndrome)

Exclusion Criteria:

* Volunteers with low levels of education (voluntary functional illiterate) that prevents the questionnaires and understanding of the guidelines made
* Working mothers of nocturnal period

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2013-08 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
sleep patterns of the study population | Baseline
  Since the mother-caregiver dedicates herself entirely to her son, we will performe overnight polysomnography to assess the sleep pattern.

SECONDARY OUTCOMES:
Hormonal profile | Baseline
  To assess the health profile of caregivers-mothers are analyzed some markers that may indicate an impairment or damage to the health of each of the parameters:
  Insulin Cortisol Luteinizing hormone (LH) Follicle-stimulating hormone (FSH) Total Testosterone Estradiol Progesterone Vitamin B12 Adrenocorticotropic hormone (ACTH)
Inflammatory profile | Baseline
  To assess the health profile of caregivers-mothers are analyzed some markers that may indicate an impairment or damage to the health of each of the parameters:
  C-reactive protein (PCR) Immunoglobulin A (IgA) Immunoglobulin G (IgG) Immunoglobulin M (IgM) Complement (C3) Complement (C4) Interleukin 6 Interleukin 10 Interleukin 1β Interleukin 2 Interleukin 4 Interleukin 8 Interferon-gamma (IFN-γ) Endothelin Prostaglandin E2 Intercellular Adhesion Molecule 1 (ICAM) Vascular cell adhesion protein 1 (VCAM) Tumor necrosis factor (TNFα) Adiponectin Leptin Cysteine Lymphocytes subpopulations (T e B)
Cardiovascular profile | Baseline
  To assess the health profile of caregivers-mothers are analyzed some markers that may indicate an impairment or damage to the health of each of the parameters:
  Homocysteine Myoglobin Cardiac troponin I Creatine kinase (CK) Creatine kinase MB (CKMB)
Metabolic profile | Baseline
  To assess the health profile of caregivers-mothers are analyzed some markers that may indicate an impairment or damage to the health of each of the parameters:
  Glucose Total cholesterol and fractions Triglycerides Uric acid Creatinine Urea Sodium Potassium Hemogram Erythrocyte sedimentation rate Natriuretic Peptide B

CONTACTS AND LOCATIONS:
Locations (1):
- University Federal of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Donders J, Taneja C. Neurobehavioral characteristics of children with Duchenne muscular dystrophy. Child Neuropsychol. 2009 May;15(3):295-304. doi: 10.1080/09297040802665777. Epub 2009 Jan 22. PMID 19160150
- [Background] Draper BM, Poulos CJ, Cole AM, Poulos RG, Ehrlich F. A comparison of caregivers for elderly stroke and dementia victims. J Am Geriatr Soc. 1992 Sep;40(9):896-901. doi: 10.1111/j.1532-5415.1992.tb01986.x. PMID 1512385
- [Background] Fee RJ, Hinton VJ. Resilience in children diagnosed with a chronic neuromuscular disorder. J Dev Behav Pediatr. 2011 Nov;32(9):644-50. doi: 10.1097/DBP.0b013e318235d614. PMID 22008789
- See also: Sleep research society — http://www.sleepresearchsociety.org/